CLINICAL TRIAL: NCT06208475
Title: The Effects of Resistance Exercise on Appetite Control, Food Reward, and Energy Intake in Different Menstrual Cycles
Brief Title: Different Menstrual Cycle in Eating Behavior Following Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202303HM002
Record Dates: First submitted 2024-01-04; First posted 2024-01-17 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Menstruation; Energy Balance; Appetitive Behavior; Food Reward
Keywords: Early follicular phase; Mid-luteal phase
MeSH Terms: conditions — Appetitive Behavior | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The exercise in the follicular phase (EF) (Experimental): Resistance exercise during the early-follicular phase (approximately during days 1-7 of the menstrual cycle).
  Interventions: Other: Resistance exercise
- The exercise in the luteal phase (EL) (Experimental): Resistance exercise during the mid-luteal phase (approximately during days 18-25 of the menstrual cycle).
  Interventions: Other: Resistance exercise
- The control in the follicular phase (CF) (No Intervention): Sit and rest during the early-follicular phase (approximately during days 1-7 of the menstrual cycle).
- The control in the luteal phase (CL) (No Intervention): Sit and rest during the mid-luteal phase (approximately during days 18-25 of the menstrual cycle).

INTERVENTIONS:
Other: Resistance exercise — Resistance exercises in the following order: squat, bench press, deadlift. Each exercise consisted of 3 sets with 7 repetitions, using a load of 70% 1RM with 120sec of rest between sets.
  Arms: The exercise in the follicular phase (EF); The exercise in the luteal phase (EL)

SUMMARY:
The study aims to provide insights into how menstrual cycle phases impact appetite responses to resistance exercise in young women. Healthy young women will participate in four trials: the exercise session in the follicular phase, the exercise session in the luteal phase, the control session in the follicular phase, and the control session in the luteal phase. Various measurements will be taken, including subjective appetite perceptions, appetite hormones, food preferences, lactate levels, estradiol levels, progesterone levels, and energy intake.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-30
* Healthy female with normal menstruation
* Weight stable for at least 6 months

Exclusion Criteria:

* Overweight (BMI > 30 kg/m^2 or body fat > 30%)
* Hypertension (> 140/90 mmHg)
* Cardiovascular disease, cancer or other chronic diseases

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Subjective appetite | 4 hours during each study intervention
  The appetite perceptions are obtained through a 0-100 mm visual analog scale. The variables assessed include perceptions of hunger (i.e., "How hungry do you feel?"), satisfaction (i.e., "How satisfied do you feel?"), fullness (i.e., "How full do you feel?"), prospective food consumption (i.e., "How much do you think you can eat?"), and nausea (i.e., "How nauseous do you feel?"), with 0 indicating "not at all" and 100 signifying "extremely.".
Change in acyl-Ghrelin | 4 hours during each study intervention
  acyl-Ghrelin in pg/mL
Change in total-Ghrelin | 4 hours during each study intervention
  total-Ghrelin in pg/mL
Change in PYY | 4 hours during each study intervention
  PYY in pg/mL
Change in active-GLP-1 | 4 hours during each study intervention
  active-GLP-1 in pg/mL
Change in total-GLP-1 | 4 hours during each study intervention
  total-GLP-1 in pg/mL
Change in lactate | 4 hours during each study intervention
  insulin in mmol/L

SECONDARY OUTCOMES:
Explicit liking | 4 hours during each study intervention
  A visual analog scale ranging from 0 to 100 mm is utilized to evaluate the question, "How pleasant would it be to taste some of this food now?" with 0 indicating "not at all" and 100 signifying "extremely."
Explicit wanting | 4 hours during each study intervention
  A visual analog scale ranging from 0 to 100 mm is utilized to evaluate the question, "How much do you want some of this food now?" with 0 indicating "not at all" and 100 signifying "extremely."
Implicit wanting | 4 hours during each study intervention
  Participants are given a set of food image pairs and are asked to select their preference by answering the question, "Which food do you desire the most at the moment?". The implicit wanting calculation involves further consideration of response time data based on preference choices using a standardized equation.
Relative preference | 4 hours during each study intervention
  Participants are given a set of food image pairs and are asked to select their preference by answering the question, "Which food do you desire the most at the moment?". The relative preference is the sum of the times each type of food is chosen, with a maximum value of 48 and a minimum value of 0.
Fat appeal bias | 4 hours during each study intervention
  Fat preference (high or low) is calculated by subtracting the mean low-fat scores from the mean high-fat scores. Positive values suggest a preference for high-fat foods, while negative scores indicate a preference for low-fat or savory foods, and a score of 0 signifies an equal preference between fat content.
Taste appeal bias | 4 hours during each study intervention
  Taste preference (savoury or sweet) is calculated by subtracting the mean savory scores from the mean sweet scores. Positive values suggest a preference for sweet foods, while negative scores indicate a preference for savory foods, and a score of 0 signifies an equal preference between taste categories.
Change in TG | 4 hours during each study intervention
  TG in mg/dL
Change in glucose | 4 hours during each study intervention
  glucose in mg/dL
Change in insulin | 4 hours during each study intervention
  insulin in mU/L
Sex hormones | 4 hours during each study intervention
  Sex hormones will be measured, such as estrogen and progesterone
Energy intake | 3 days during each study intervention
  Participants will be required to record their diet for the day before, the current day, and the day following the experiment.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Wen Liu, Ph.D., Principal Investigator — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No